CLINICAL TRIAL: NCT01164683
Title: A Pilot Study of CPAP Adherence Promotion by Peer Buddies With Sleep Apnea
Acronym: CPAPPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPO 10-066
Record Dates: First submitted 2010-06-15; First posted 2010-07-19 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2013-02

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; adherence
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Trained peers with sleep apnea will be paired with the newly diagnosed patients over a 3-month period. During this time the trained peers will share experiences on coping strategies with CPAP device and equipment (promote self efficacy), share their positive experiences (motivational effects and outcome expectancies), share their knowledge of perceived vulnerabilities due to untreated sleep apnea (promote risk perception), share methods for improving efficacy of CPAP equipment and interface (patient education) and prepare their subjects for upcoming physician or respiratory therapist appointments (patient activation).
  Interventions: Behavioral: Peer-driven intervention
- Arm 2 (Active Comparator): Usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Peer-driven intervention — Trained peers with sleep apnea will be paired with the newly diagnosed patients over a 3-month period. During this time the trained peers will share experiences on coping strategies with CPAP device and equipment (promote self efficacy), share their positive experiences (motivational effects and outcome expectancies), share their knowledge of perceived vulnerabilities due to untreated sleep apnea (promote risk perception), share methods for improving efficacy of CPAP equipment and interface (patient education) and prepare their subjects for upcoming physician or respiratory therapist appointments (patient activation).
  Other Names: Peer-buddy system (PBS)
  Arms: Arm 1
Other: Usual Care — All participants will receive usual care following initiation of CPAP therapy. Visits with respiratory therapist and sleep physician wherein patients are educated about the basics of the care and operation of the device, mask and related equipment. Subsequently, their CPAP adherence is monitored and appropriate interventions such as mask change and re-education undertaken as needed.
  Arms: Arm 2

SUMMARY:
Obstructive sleep apnea (OSA) is a highly prevalent condition in veterans with some estimates as high as 47%. Poor adherence to the primary treatment of OSA -- continuous positive airway pressure (CPAP) therapy - is associated with increased risk for heart attacks, strokes and even death. The investigators plan to improve CPAP adherence in veterans through their interactions with peers who have successfully adopted CPAP therapy.

Such "peer-buddies" may promote the well-being of veterans while remaining highly cost-effective when compared to healthcare providers. Our strategy is grounded on the rationale that veterans as a group are ecoculturally more homogenous than expected for the given level of differences in age, gender, ethnicity, or socioeconomic strata. Our long-term objectives are to initiate a larger, multi-site, research study for enhancing CPAP adherence in veterans with OSA. The ultimate goal of this research is to develop a cheap, effective and exportable system of care to promote CPAP adherence in patients with OSA.

DETAILED DESCRIPTION:
Project background: Obstructive sleep apnea (OSA) is a prevalent condition that is most frequently treated with continuous positive airway pressure (CPAP) therapy. Non-adherence to such therapy, however, afflicts a high proportion of adults with sleep apnea (46-83%). Moreover, such non-adherence to CPAP is associated with increased risk for fatal and non-fatal cardiovascular events. There remains a paucity of reliable and cost-effective interventions that could promote CPAP adherence. Promoting adherence to therapy through peer-driven intervention is cheap and has met with modest success in other chronic conditions such as HIV, heart failure and diabetes mellitus. Whether such a peer-driven ("buddy") system can improve adherence to CPAP therapy is unknown.

Project Objectives: Our overall aim is to assess the feasibility and acceptability of a CPAP adherence program driven by trained "peer-buddies" with sleep apnea. Specific Objective #1: To evaluate patient ratings of the acceptability of the peer buddy system (PBS) in veterans receiving CPAP therapy for OSA. Specific Objective #2: To obtain preliminary data on the effectiveness of PBS on sleep-specific HR-QOL (Functional outcomes in sleep questionnaire [FOSQ]) in veterans receiving CPAP therapy for OSA. Specific Objective #3: To obtain preliminary data on the effect of PBS on CPAP adherence, vigilance, patient activation, and self-efficacy in veterans receiving CPAP therapy for OSA.

Project Methods: In order to address these aims, we will recruit recently diagnosed patients with OSA who have not been initiated on CPAP therapy and randomly assign them to the peer-buddy system to promote adherence to CPAP therapy (intervention group) or be assigned to usual care (control group). In the PBS intervention group, trained peers with sleep apnea will be paired with the newly diagnosed patients over a 3- month period. During this time the trained peers will share experiences on coping strategies with CPAP device and equipment (promote self efficacy), share their positive experiences (motivational effects and outcome expectancies), share their knowledge of perceived vulnerabilities due to untreated sleep apnea (promote risk perception), share methods for improving efficacy of CPAP equipment and interface (patient education) and prepare their subjects for upcoming physician or respiratory therapist appointments (patient activation). The interaction will occur during supervised "in-person" sessions and during telephonic conversations over the 3-month period. Subjects from both groups will be reassessed at the end of 3 months in order to determine objective measures of CPAP adherence, sleep-specific HRQOL Functional outcomes of sleep questionnaire [FOSQ]), vigilance (psychomotor vigilance testing), measures of self-efficacy (outcome expectancy, treatment self-efficacy, and risk perception [SEMSA questionnaire]) and patient activation (Patient Activation Measure [PAM]).

ELIGIBILITY:
Inclusion Criteria:

1. Obstructive Sleep Apnea (defined by Apnea-hypopnea index [AHI] > 5 per hour; with hypopneas defined as greater than 30% reduction in airflow with 4 or greater drop in oxygen saturation). AHI will be determined by full night or split-night polysomnography.
2. Age range 21 - 85 years old.
3. Stable medical history and no change in medications, including anti-hypertensive and thyroid replacement, in the previous 4 months.
4. No regular use (> 3 times/week) of sedative or hypnotic medications in the last 4 months.

Exclusion Criteria:

1. Central sleep apnea (central apnea index > 5 per hour and >50% of Apnea-hypopnea index constituted by central apneas and non-obstructive hypopneas).
2. Complex sleep apnea or CPAP emergent central apnea (Central apnea index > 5 per hour during CPAP titration with >50% of Apnea-hypopnea index constituted by central apneas and non-obstructive hypopneas).
3. Requiring oxygen or bi-level positive airway pressure for treatment of OSA or hypoventilation.
4. Decompensated cardiac (heart failure or angina) or pulmonary (severe COPD or uncontrolled asthma) disease
5. Chronic narcotic use
6. Nasal obstruction (nasal congestion score > 15) or enlarged tonsils
7. Diagnosis of another sleep disorder in addition to OSA based on PSG (e.g., periodic limb movement disorder [ 15 limb movements/hour of sleep with arousal], central sleep apnea [ 50% of apneas on diagnostic PSG are central apneas], insomnia, obesity hypoventilation syndrome, or narcolepsy).
8. Previous treatment with positive airway pressure, home oxygen therapy, tracheotomy, uvulopalatopharyngoplasty, or other surgery for OSA.
9. Night shift workers in situations or occupations where they regularly experience jet lag, or have irregular work schedules by history over the last 6 months.
10. Routine consumption of more than 2 alcoholic beverages per day.
11. Recent or recurring history of recreational drug use leading to tolerance or dependence.
12. Unable to perform tests due to inability to communicate verbally, inability to write and read in English; less than a 5th grade reading level; visual, hearing or cognitive impairment (e.g. previous head injury); or upper extremity motor deficit (e.g., previous stroke that prevents patient from using CPAP treatment).

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Functional Outcomes of Sleep Questionnaire (FOSQ) | Three months

SECONDARY OUTCOMES:
CPAP adherence | Three months
Patient Activation Measure (PAM) survey assessment tool | Three months
Self efficacy measure for sleep apnea | Three months
Psychomotor vigilance test | three months
Patient acceptability of peer-based intervention | Three months
Epworth sleepiness score | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Sairam Parthasarathy, MD, Principal Investigator — Southern Arizona VA Health Care System, Tucson, AZ
Locations (1):
- Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona, United States

REFERENCES:
- [Background] Parthasarathy S. The need for pharmacovigilance in sleep medicine. Sleep. 2011 Jul 1;34(7):827-8. doi: 10.5665/SLEEP.1096. No abstract available. PMID 21731126
- [Derived] Parthasarathy S, Wendel C, Haynes PL, Atwood C, Kuna S. A pilot study of CPAP adherence promotion by peer buddies with sleep apnea. J Clin Sleep Med. 2013 Jun 15;9(6):543-50. doi: 10.5664/jcsm.2744. PMID 23772186